CLINICAL TRIAL: NCT06201741
Title: A Study to Evaluate the Human Biodistribution and Dosimetry of the Radionuclide Labeled ZT-111 in Patients With Metastatic Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-1018
Record Dates: First submitted 2024-01-02; First posted 2024-01-11 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Prostate Specific Membrane Antigen Positive Metastatic Prostate Cancer
Keywords: PSMA positive metastatic prostate cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- [131I]/[18F]/[68Ga]ZT-111 (Experimental): [131I]/[18F]/[68Ga]ZT-111, single dose
  Interventions: Radiation: [131I]/[18F]/[68Ga]ZT-111

INTERVENTIONS:
Radiation: [131I]/[18F]/[68Ga]ZT-111 — [131I]/[18F]/[68Ga]ZT-111, single dose

SUMMARY:
This study is to evaluate the safety, biodistribution, radiation dosimetry and tumor uptake of the [131I]/[18F]/[68Ga]ZT-111 in patients with PSMA positive metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 65 years old.
2. Histologically or cytologically confirmed prostate adenocarcinoma with documented history of ≥1 metastatic lesions indicated by imaging.
3. Informed consent must be obtained in writing from the subject, their legally authorized representative, or caregiver.
4. Willing and able to comply with all aspects of this study.

Exclusion Criteria:

1. Severe hepatic or renal impairment.
2. History of major surgery within the last month.
3. Participation in another concurrent clinical trial.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2023-12-27 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Dosimetry | About 24hours from time of injection
  Whole body and organ uptake activity

SECONDARY OUTCOMES:
Incidence and severity of adverse events | From administration of [131I]/[18F]/[68Ga]ZT-111 until 1 week after injection
  Incidence and severity of adverse events (AEs) as assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided